CLINICAL TRIAL: NCT04033835
Title: Mentalization Based Treatment - Introductory Group for Male Prisoners With Borderline and/or Antisocial Personality Disorder in Her Majesty's Prison Barlinnie
Brief Title: Mentalization Based Treatment - Introductory (MBT-I) Group for Male Prisoners With Borderline and/or Antisocial Personality Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: GN19MH314
Record Dates: First submitted 2019-07-10; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Borderline Personality Disorder (BPD); Antisocial Personality Disorder (ASPD)
MeSH Terms: conditions — Borderline Personality Disorder; Antisocial Personality Disorder | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBT-I (Experimental): 12 sessions of MBT
  Interventions: Other: Mentalization Based Treatment-Introductory
- Waiting list control (Active Comparator): Treatment as usual
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Mentalization Based Treatment-Introductory — Mentalization Based Treatment-Introductory
  Arms: MBT-I
Other: Treatment as usual — Treatment as usual
  Arms: Waiting list control

SUMMARY:
Established evidence base with MBT for treatment of Borderline Personality Disorder (BPD) and/or Antisocial Personality Disorder (ASPD). Demographic information of United Kingdom prison population highlights large proportion of offenders with PD. There is no agreed universal approach to treatment of PD within Scottish prisons with large variance across the prison estate. MBT pilots in HMP Edinburgh and HMP Cornton Vale have demonstrated positive findings in female offenders which could be replicated in male populations.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of BPD and/or ASPD
* Co-morbidity with other personality disorder is accepted
* Sentenced prisoners with estimated date of liberation > six months

Exclusion Criteria:

* Co-morbid severe and enduring mental illness (schizophrenia, delusional disorder, bipolar affective disorder, major depressive disorder)
* Co-morbid organic brain disorder (acquired brain injury, alcohol related brain damage)
* Remand prisoners
* Uncontrolled substance dependence
* Index offence of sexual offending
* Repeatedly chaotic, antisocial or violent behaviour in prison
* Care in segregation and reintegration unit in past 3 months
* Current individual specialist psychological therapy in prison
* English as not first language

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Completion of three MBT-I group cycles | 18 months
  Participants to have attended ≥75% (9 or more out of 12) of scheduled sessions to consider this successful completion of the programme.
  ≥50% participants who commenced session one to have completed the intervention as described above to consider the group successful.

SECONDARY OUTCOMES:
Quantitative data measuring change in difficulties with interpersonal relationships pre- and post-intervention | 21 months
  Inventory of Interpersonal Problems-32 (IIP-32) to be administered one week pre-, one week post- and three months post-intervention. The scale measures difficulties with interpersonal relationships which are a core feature of personality disorder psychopathology.
  There are 32 items scored on a 5 point scale (0-4) measuring 2 domains of affiliating and distancing (16 items each) difficulties with interpersonal relationships. There are 8 differing interpersonal relationship styles (4 each for affiliating and distancing). The maximum score therefore for each style is 16 (4 x 4 point scores), for each domain is 64 (16 x 4 point scores), and total score is 128 (32 x 4 point scores). The minimum score is 0. Higher values indicate increasing severity.
Quantitative data measuring change in difficulties with interpersonal relationships pre- and post-control | 21 months
  Inventory of Interpersonal Problems-32 (IIP-32) to be administered one week pre-, one week post- and three months post-intervention. The scale measures difficulties with interpersonal relationships which are a core feature of personality disorder psychopathology.
  There are 32 items scored on a 5 point scale (0-4) measuring 2 domains of affiliating and distancing (16 items each) difficulties with interpersonal relationships. There are 8 differing interpersonal relationship styles (4 each for affiliating and distancing). The maximum score therefore for each style is 16 (4 x 4 point scores), for each domain is 64 (16 x 4 point scores), and total score is 128 (32 x 4 point scores). The minimum score is 0. Higher values indicate increasing severity.
Quantitative data measuring change in difficulties with impulsivity pre- and post-intervention | 21 months
  Barrett Impulsiveness Scale (BIS) to be administered one week pre-, one week post- and three months post-intervention. The scale measures difficulties with impulsivity which is a core feature of personality disorder psychopathology.
  There are 30 items scored on a 4 point (1-4) scale measuring impulsivity. The maximum score is 120 (30 x 4 point scores). The minimum score is 30 (30 x 1 point scores). Higher values indicate increasing severity.
Quantitative data measuring change in difficulties with impulsivity pre- and post-control | 21 months
  Barrett Impulsiveness Scale (BIS) to be administered one week pre-, one week post- and three months post-intervention. The scale measures difficulties with impulsivity which is a core feature of personality disorder psychopathology.
  There are 30 items scored on a 4 point (1-4) scale measuring impulsivity. The maximum score is 120 (30 x 4 point scores). The minimum score is 30 (30 x 1 point scores). Higher values indicate increasing severity.
Quantitative data measuring change in difficulties with reflective functioning pre- and post-intervention | 21 months
  Reflective Functioning Questionnaire (RFQ) to be administered one week pre-, one week post- and three months post-intervention. The scale measures difficulties with reflective functioning which is a core feature of personality disorder psychopathology.
  There are 54 items scored on a 7 point (1-7) scale measuring 2 domains of certainty and uncertainty (26 items each) difficulties with reflective functioning. Two items do not score. Only extreme rankings score points for each item (i.e 7 or 1 scores 3, 6 or 2 scores 2 and 5 or 3 scores 1 depending on the item type). The maximum score therefore for each domain is 78 (26 x 3 point scores), and total score is 156 (52 x 3 point scores). The minimum score is 0. Higher values indicate increasing severity.
Quantitative data measuring change in difficulties with reflective functioning pre- and post-control | 21 months
  Reflective Functioning Questionnaire (RFQ) to be administered one week pre-, one week post- and three months post-intervention. The scale measures difficulties with reflective functioning which is a core feature of personality disorder psychopathology.
  There are 54 items scored on a 7 point (1-7) scale measuring 2 domains of certainty and uncertainty (26 items each) difficulties with reflective functioning. Two items do not score. Only extreme rankings score points for each item (i.e 7 or 1 scores 3, 6 or 2 scores 2 and 5 or 3 scores 1 depending on the item type). The maximum score therefore for each domain is 78 (26 x 3 point scores), and total score is 156 (52 x 3 point scores). The minimum score is 0. Higher values indicate increasing severity.
Quantitative data measuring change in depressive symptoms pre- and post-intervention | 21 months
  Beck's Depression Inventory (BDI) to be administered one week pre-, one week post- and three months post-intervention. The scale measures depressive symptoms which are a common feature of personality disorder psychopathology.
  There are 21 items scored on a 4 point (0-3) scale measuring depressive symptoms. The maximum score is 63 (21 x 3 point scores). The minimum score is 0. Higher values indicate increasing severity (1-10 - these ups and downs are considered normal; 11-16 - mild mood disturbance; 17-20 - borderline clinical depression; 21-30 - moderate depression; 31-40 - severe depression; >40 - extreme depression).
Quantitative data measuring change in depressive symptoms pre- and post-control | 21 months
  Beck's Depression Inventory (BDI) to be administered one week pre-, one week post- and three months post-intervention. The scale measures depressive symptoms which are a common feature of personality disorder psychopathology.
  There are 21 items scored on a 4 point (0-3) scale measuring depressive symptoms. The maximum score is 63 (21 x 3 point scores). The minimum score is 0. Higher values indicate increasing severity (1-10 - these ups and downs are considered normal; 11-16 - mild mood disturbance; 17-20 - borderline clinical depression; 21-30 - moderate depression; 31-40 - severe depression; >40 - extreme depression).
Quantitative data measuring change in anxiety symptoms pre- and post-intervention | 21 months
  Beck's Anxiety Inventory (BAI) to be administered one week pre-, one week post- and three months post-intervention. The scale measures anxiety symptoms which are a common feature of personality disorder psychopathology.
  There are 21 items scored on a 4 point (0-3) scale measuring anxiety symptoms. The maximum score is 63 (21 x 3 point scores). The minimum score is 0. Higher values indicate increasing severity (0-21 - low anxiety; 22-35 - moderate anxiety; >35 - potentially concerning levels of anxiety).
Quantitative data measuring change in anxiety symptoms pre- and post-control | 21 months
  Beck's Anxiety Inventory (BAI) to be administered one week pre-, one week post- and three months post-intervention. The scale measures anxiety symptoms which are a common feature of personality disorder psychopathology.
  There are 21 items scored on a 4 point (0-3) scale measuring anxiety symptoms. The maximum score is 63 (21 x 3 point scores). The minimum score is 0. Higher values indicate increasing severity (0-21 - low anxiety; 22-35 - moderate anxiety; >35 - potentially concerning levels of anxiety).
Quantitative data measuring change in social functioning and satisfaction pre- and post-intervention | 21 months
  Social Adjustment Scale - Self Report (SAS-SR) to be administered one week pre-, one week post- and three months post-intervention. The scale measures difficulties with social functioning and satisfaction which are common sequelae of personality disorder.
  There are 54 items scored measuring instrumental and expressive performance over the past two weeks. They examine across 6 domains - work, social and leisure, extended family, primary relationship, parental, family unit. Within these domains, the items cover 4 categories - performance, friction with people, finer aspects of interpersonal relations, and feelings and satisfactions.
Quantitative data measuring change in social functioning and satisfaction pre- and post-control | 21 months
  Social Adjustment Scale - Self Report (SAS-SR) to be administered one week pre-, one week post- and three months post-intervention. The scale measures difficulties with social functioning and satisfaction which are common sequelae of personality disorder.
  There are 54 items scored measuring instrumental and expressive performance over the past two weeks. They examine across 6 domains - work, social and leisure, extended family, primary relationship, parental, family unit. Within these domains, the items cover 4 categories - performance, friction with people, finer aspects of interpersonal relations, and feelings and satisfactions.
Quantitative data measuring change in overall symptoms and functioning pre- and post-intervention | 21 months
  Clinical Outcomes in Routine Evaluation - Outcome Measure (CORE-OM) to be administered one week pre-, one week post- and three months post-intervention. The scale measures overall change in symptoms and functioning from baseline following completion of the intervention.
  There are 34 items scored on a 5 point (0-4) scale measuring overall change across 4 domains - subjective well-being (4 items), problems and symptoms (12 items), life functioning (12 items), and risk and harm (6 items). The maximum score is 136 (34 x 4 point scores). The minimum score is 0. Higher values indicate increasing severity.
Quantitative data measuring change in overall symptoms and functioning pre- and post-control | 21 months
  Clinical Outcomes in Routine Evaluation - Outcome Measure (CORE-OM) to be administered one week pre-, one week post- and three months post-intervention. The scale measures overall change in symptoms and functioning from baseline following completion of the intervention.
  There are 34 items scored on a 5 point (0-4) scale measuring overall change across 4 domains - subjective well-being (4 items), problems and symptoms (12 items), life functioning (12 items), and risk and harm (6 items). The maximum score is 136 (34 x 4 point scores). The minimum score is 0. Higher values indicate increasing severity.
Quantitative data from behavioural proxy measures examining change in the number of challenging behaviours pre- and post-intervention | 21 months
  The number of discipline procedures (reports) and Incentives and Enhanced Privileges (IEPs) will be examined over a three month period pre-intervention, three month period during the intervention and three month period post-intervention. This allows a behavioural proxy measure of negative (reports) vs. positive (IEPs) behaviours.
Quantitative data from behavioural proxy measures examining change in the number of challenging behaviours pre- and post-control | 21 months
  The number of discipline procedures (reports) and Incentives and Enhanced Privileges (IEPs) will be examined over a three month period pre-intervention, three month period during the intervention and three month period post-intervention. This allows a behavioural proxy measure of negative (reports) vs. positive (IEPs) behaviours.
Qualitative data from follow up interviews of participants examining understanding of and overall satisfaction of intervention | 21 months
  Semi-structured interview schedule to be completed one week post- and three months post- intervention. This will examine participant's understanding of the concepts of the intervention, in addition to their overall satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No